CLINICAL TRIAL: NCT04024371
Title: Validating Reward-related Biomarkers to Facilitate Development of New Treatments for Anhedonia and Reward Processing Deficits in Schizophrenia and Major Depressive Disorder
Brief Title: Validating Reward-related Biomarkers (RTOC)
Acronym: RTOC
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Collaborators: P1vital Products LTD. (Unknown); Biotrial (Industry); University Hospital Frankfurt, Department of Psychiatry, Psychosomatic Medicine and Psychotherapy (Unknown); The Institute of Neuropsychiatry and Addictions (INAD), Parc de Salut Mar, Barcelona (Unknown); Aristotle University Of Thessaloniki (Other); Maastricht University, School for Mental Health and Neuroscience (Unknown)
Responsible Party: Sponsor
Other Study IDs: RTOC1
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Schizophrenia; Depression; Motivation; Anhedonia, Physical; Anhedonia, Social; Negative Symptoms With Primary Psychotic Disorder
MeSH Terms: conditions — Schizophrenia; Depression; Anhedonia | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HV: Humans aged 20-55 without a diagnosis of a psychiatric and neurological disorder.
  Interventions: Behavioral: Self-rating Questionnaires; Behavioral: Measures of Reward processing/reinforcement learning
- SZ: Humans aged 20-55 with a primary Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) diagnosis of Schizophrenia.
  Interventions: Behavioral: Self-rating Questionnaires; Behavioral: Measures of Reward processing/reinforcement learning; Behavioral: Additional Schizophrenia-specific Questionnaires and Interviews
- MDD: Humans aged 20-55 with a primary Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) diagnosis of MDD.
  Interventions: Behavioral: Self-rating Questionnaires; Behavioral: Measures of Reward processing/reinforcement learning

INTERVENTIONS:
Behavioral: Self-rating Questionnaires — * Snaith-Hamilton Pleasure Scale (SHAPS; Snaith et al. 1995)
  * Quick Inventory of Depressive Symptomatology (QIDS; 16 items)
  * Behavioral avoidance/inhibition Scales (BIS/BAS)
Behavioral: Measures of Reward processing/reinforcement learning — * Grip Strength Effort Task (Reddy et al. 2015; in combination with EEG)
  * Doors (Gambling) task (Foti and Hajcak 2009; in combination with EEG)
  * Reinforcement Learning/Working Memory task (Collins et al. 2017; no EEG)
Behavioral: Additional Schizophrenia-specific Questionnaires and Interviews — * Positive and Negative Syndrome Scale (PANSS: Kay et al. 1987)
  * Brief Negative Symptom Scale (BNSS; Kirkpatrick et al. 2011)
  Groups: SZ

SUMMARY:
Deficits or abnormalities in reward processing are present in a number of psychiatric disorders. The overarching objective of the study is to conduct initial validation work towards optimising three experimental tasks - which have previously been shown to be sensitive to reward processing deficits - for future use in clinical trials.

This initial validation work has the primary objective to uncover group differences in task outcome measures between healthy control participants, participants with Major Depressive Disorder (MDD) and participants with schizophrenia (SZ) using statistical analyses. This may provide some indications for the use of these tasks as clinically-relevant biomarkers.

Primary aims include:

(i) comparing the investigator's endpoint means and distributions to those in previously published data; (ii) replication of previously-reported differences between MDD/SZ vs. healthy control participants, and, (iii) exploring the relationship between task endpoints and subjective participant- and clinician-rated report of reward-related constructs (e.g. anhedonia, negative symptoms).

ELIGIBILITY:
General:

1. Be able to provide signed and dated informed consent for study participation.
2. Be male or female, aged between 20 and 55 years, inclusive.
3. Be able to read, write, and speak the language in which psychometric tests are provided, with acceptable visual and auditory acuity (corrected if necessary).
4. Unless otherwise stated, CNS medications to treat symptoms of MDD or SZ and other stable CNS conditions requiring medication is permitted in the MDD and SZ groups, provided the daily dose of medication has not been changed by more than +/- 30% in the last 4 weeks before the start of the study, and is not expected to change by a larger fraction while participating in the study.

MDD

Participants must:

1. Have a primary Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) diagnosis of MDD, confirmed by the result of the MINI interview conducted by the site at screening. Subjects with a diagnosis of comorbid Generalized Anxiety Disorder (GAD), Social Anxiety Disorder (SAD), Panic Disorder or specific phobia may be included.
2. Meet the DSM-5 criteria for a current Major Depressive Episode, with the current depressive episode not having lasted longer than 6 months.
3. If undergoing treatment, be currently treated with an antidepressant approved in this protocol for at least 4 continuous weeks. Psychological treatments (e.g., Cognitive Behaviour Therapy, Interpersonal Psychotherapy, Psychodynamic Psychotherapy etc.) are all permitted in this study regardless of frequency and duration.

SZ

Subjects must:

1. Have a primary diagnosis of schizophrenia according to the Statistical Manual of Mental Disorders 5th edition (DSM-5), confirmed by the result of the MINI interview conducted by the site at screening. Subjects with a diagnosis of comorbid Generalized Anxiety Disorder (GAD), Social Anxiety Disorder (SAD), Panic Disorder or specific phobia may be included.
2. Dose of antipsychotics not exceeding the equivalent of 6 mg risperidone.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A sample of 37 completed individuals with MDD, 37 completed individuals with SZ, and a maximum of 80 healthy volunteers (without a neurological or psychiatric disorder) who will not differ on age or gender.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Grip effort outcome | Day 1
  Percentage of hard task choices at different reward levels
Doors task outcome | Day 1
  "Feedback negativity", an event-related potential (ERP) at approximately 300ms after feedback presentation indicating a favourable versus unfavourable outcome in paradigms in which the participant loses or wins money.
RL/WM task outcome | Day 1
  Accuracy as function of set size (difficulty)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hernaus, PhD, Study Director — Maastricht University
Locations (4):
- University Hospital Frankfurt, Department of Psychiatry, Psychosomatic Medicine and Psychotherap, Frankfurt, Germany
- Aristotle University of Thessaloniki, School of Medicine, Department of Clinical Pharmacology, Thessaloniki, Greece
- Maastricht University, Maastricht, Netherlands
- Institute of Neuropsychiatry and Addictions (INAD), Parc de Salut Mar, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The RTOC clinical study has received funding from Boehringer Ingelheim International GmbH, H. Lundbeck, Janssen Pharmaceutica, Blackthorn Therapeutics, and F. Hoffmann-La Roche Ltd. All individual data will be made available to these parties.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Background] Foti D, Hajcak G. Depression and reduced sensitivity to non-rewards versus rewards: Evidence from event-related potentials. Biol Psychol. 2009 Apr;81(1):1-8. doi: 10.1016/j.biopsycho.2008.12.004. Epub 2008 Dec 31. PMID 19162124
- [Background] Collins AGE, Albrecht MA, Waltz JA, Gold JM, Frank MJ. Interactions Among Working Memory, Reinforcement Learning, and Effort in Value-Based Choice: A New Paradigm and Selective Deficits in Schizophrenia. Biol Psychiatry. 2017 Sep 15;82(6):431-439. doi: 10.1016/j.biopsych.2017.05.017. Epub 2017 May 31. PMID 28651789
- [Result] Reddy LF, Horan WP, Barch DM, Buchanan RW, Dunayevich E, Gold JM, Lyons N, Marder SR, Treadway MT, Wynn JK, Young JW, Green MF. Effort-Based Decision-Making Paradigms for Clinical Trials in Schizophrenia: Part 1-Psychometric Characteristics of 5 Paradigms. Schizophr Bull. 2015 Sep;41(5):1045-54. doi: 10.1093/schbul/sbv089. Epub 2015 Jul 3. PMID 26142081
- [Derived] Bilderbeck AC, Raslescu A, Hernaus D, Hayen A, Umbricht D, Pemberton D, Tiller J, Sogaard B, Sambeth A, van Amelsvoort T, Reif A, Papazisis G, Perez V, Elices M, Maurice D, Bertaina-Anglade V, Dawson GR, Pollentier S. Optimizing Behavioral Paradigms to Facilitate Development of New Treatments for Anhedonia and Reward Processing Deficits in Schizophrenia and Major Depressive Disorder: Study Protocol. Front Psychiatry. 2020 Nov 5;11:536112. doi: 10.3389/fpsyt.2020.536112. eCollection 2020. PMID 33250788